CLINICAL TRIAL: NCT03337880
Title: Neonatal Outcomes in Instrumental Delivery: Newborn Head Mark and Comfort.
Brief Title: Neonatal Outcomes in Instrumental Delivery
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CNEI
Record Dates: First submitted 2017-11-06; First posted 2017-11-09 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2017-12

CONDITIONS: Instrumental Delivery; Nec, Affecting Fetus or Newborn
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: newborns who were delivered with an extractor
  Interventions: Other: instrumental delivery
- Controls: newborns who were not delivered with an extractor

INTERVENTIONS:
Other: instrumental delivery — the birth was assisted with an extractor.
  Groups: Cases

SUMMARY:
The aim of this study is to compare the impact of instrumental delivery on newborn head mark and newborn comfort over the impact of non-instrumental delivery. It is also to evaluate how mothers age, Body Mass Index, instrumental extraction indication, extractor type, variety and height of the fetal presentation, operator, time of birth (day or night) and birth weight impact on head mark existence and newborn comfort.

ELIGIBILITY:
Inclusion Criteria:

* term infant
* non-opposition of the newborn parent

Exclusion Criteria:

* outborn child
* premature newborn
* newborn transferred

Ages: 12 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: mature newborns who profit an instrumental delivery or not.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Head mark or injury | 12 to 72 hours of age
  Any mark or injury (skin erosion, wound, hematoma, fracture, paralysis, etc.) on the newborn head will be described (type, color, size, position) and documented (photo)
Newborn comfort | 12 to 72 hours of age
  assessed using Newborn Pain and Discomfort Scale (EDIN) (DEBILLON et al. Development and initial validation of the EDIN scale, a new tool for assessing prolonged pain in preterm infants. Arch Dis Child Neonatal Ed 2001;85:36-41)

SECONDARY OUTCOMES:
Analgesic use | 0 to 72 hours of age
  Any analgesic administration to the newborn will be reported
Length of hospitalisation after childbirth | First month of life
  The day out for home of the newborn will be reported

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers University Hospital, Poitiers, France